CLINICAL TRIAL: NCT06264531
Title: Evaluation of the Efficacy and Safety of Anti-angiogenic Therapy With Intravenous Bevacizumab in Patients With Symptomatic Cerebral Arteriovenous Malformations
Brief Title: Efficacy and Safety of Anti-angiogenic Therapy With IV Bevacizumab in Patients With Symptomatic Cerebral Arteriovenous Malformations
Acronym: BevacizuMAV
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JDS_2023_12
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Cerebral AV Malformation
MeSH Terms: conditions — Intracranial Arteriovenous Malformations | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bevacizumab (Experimental): Bevacizumab 5 mg/kg as a slow infusion over 90 minutes every 14 days for a total of 6 injections
  Interventions: Drug: Bevacizumab
- placebo (Placebo Comparator): NaCl 0.9% as a slow infusion over 90 minutes every 14 days for a total of 6 injections
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 5 mg/kg as a slow infusion over 90 minutes every 14 days for a total of 6 injections
  Arms: bevacizumab
Drug: Placebo — NaCl 0.9% slow infusion over 90 minutes every 14 days for a total of 6 injections
  Arms: placebo

SUMMARY:
Brain arteriovenous malformations (AVMs) are responsible for hemorrhagic strokes, particularly in children and young adults. They can also be responsible for chronic neurological disorders: motor or sensory deficits, disturbances of higher functions, epilepsy or disabling headaches. The management of brain AVMs is complex and requires a multidisciplinary approach in an expert center. Available therapies include endovascular embolization, neurosurgical resection and/or radiosurgery. These procedures carry a risk of neurological complications, and are reserved for small AVMs located at a distance from highly functional cerebral structures. To date, no drug therapy is recommended if interventional treatment is not possible.

Several studies on resected brain AVM tissue have demonstrated that these malformations are the site of significant evolutionary inflammatory and neo-angiogenesis processes. Other studies have specifically shown that VEGF (vascular endothelial growth factor) levels are increased in AVMs. More recently, a pre-clinical study showed that anti-angiogenic treatment with Bevacizumab reduced vascular proliferation within AVMs in mice. Finally, a Phase II clinical trial in patients with Rendu-Osler disease (a genetic vascular disorder characterized by recurrent epistaxis, cutaneous telangiectasia and the presence of visceral AVMs) showed a clinical benefit of IV Bevacizumab on the symptomatology of these vascular malformations, with a reduction in the risk of hemorrhage and the extent of hepatic arteriovenous shunts. A randomized Phase III trial is currently underway (NCT03227263) to assess the efficacy of IV Bevacizumab in Rendu-Osler disease.

The aim of our study is to assess the efficacy of IV Bevacizumab on the disabling symptoms associated with symptomatic brain AVMs.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* With a symptomatic cerebral AVM (chronic headache, focal neurological deficit, cognitive impairment, epilepsy) of Spetzler and Martin grade III, IV or V.
* Whose symptoms are sufficiently severe to allow significant improvement with treatment:

  * MoCA score ≤ 25 and/or
  * NIHSS score ≥ 4 and/or
  * Epilepsy Balance Score ≥ 2 and/or
  * HIT-6 score ≥ 48
* With functional signs and symptoms not sequellar to a previous bleeding episode AND disabling (mRS>1)
* Ineligible for therapeutic intervention (endovascular or neurosurgery or radiosurgery)
* With normal bone marrow, liver and kidney function
* For women of childbearing potential: negative pregnancy test within 14 days of inclusion and effective contraception for up to 6 months after the end of treatment
* Having received informed consent to participate in the study
* Affiliated or beneficiary of a social security scheme

Exclusion Criteria:

* Known allergy to bevacizumab or an excipient.
* Hypersensitivity to Chinese hamster ovary (CHO) cell products or other recombinant human or humanized antibodies.
* Contraindication to cerebral MRI
* Absolute or relative contraindication to gadolinium injection
* Proteinuria ≥ 2+ on urine dipstick (patients with proteinuria ≥2+ on urine dipstick will need to have proteinuria ≤ 1g protein on 24-hour urine to be eligible)
* Uncontrolled hypertension (PAS >150 and/or PAD > 100 mmHg)
* History of hypertensive crisis or hypertensive encephalopathy
* Congestive heart failure (New York Heart Association Grade II or higher)
* Previous myocardial infarction or unstable angina in the preceding 12 months
* Symptomatic peripheral vascular disease
* Vascular disease (aortic aneurysm, aortic dissection)
* Major surgery, open biopsy or major traumatic lesion within 4 weeks prior to inclusion, or anticipation of the need for major surgery during the study.
* Biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to inclusion
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess in the 6 months prior to inclusion
* Significant unhealed wound, ulcer or bone fracture
* Thrombotic episode within 6 months prior to inclusion
* Atrial fibrillation
* Patient under legal protection
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients showing at least one of the following improvements : cognition, neurological symptoms, epilepsy symptoms, headaches. | month 6
  Proportion of patients showing at least one of the following improvements :
  * change of at least 5 points in Montreal Cognitive Assessment score (from 0 to 30 ; higher score meaning a better outcome)
  * change of at least 4 points in National Institutes of Health Stroke Scale ( from 0 to 42 : higher score meaning a worse outcome)
  * change of at least one stage on the Epilepsy Balance Score (from 1 to 5 ; higher score meaning a worse outcome)
  * change of at least 12 points on the Headache ImpactTest-6 score (from 36 to 78 : higher score meaning a worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- HFAR, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No